CLINICAL TRIAL: NCT06201637
Title: Investigation Of The Validity And Reliability Of The Short Physical Performance Battery In Patients Undergoing Total Knee Arthroplasty
Brief Title: Validity And Reliability Of The Short Physical Performance Battery In Patients Undergoing Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Damla Ozcan, Msc. Pt, Dokuz Eylul University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 6784-GOA
Record Dates: First submitted 2024-01-02; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Knee Osteoarthritis
Keywords: Total knee arthroplasty, knee, Short Physical Performance Battery, validity, reliability
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Performance Test — Performance Test

SUMMARY:
Objectives: Practical, applicable, valid, and reliable tools are needed to assess physical performance in patients with Total Knee Arthroplasty(TKA) in a variety of settings, including routine clinical assessment, research studies, and community-based programs. Therefore, the aim of this study is to evaluate the validity and reliability of the Short Physical Performance Battery (SPPB) among patients with TKA.

Methods: We included patients who underwent TKA surgery. The SPPB, Timed up and go(TUG) test and, Hospital for Special Surgery (HSS) Knee Score were administered to the patients. SPPB was performed twice on the same day with 1 h rest.

ELIGIBILITY:
Inclusion Criteria:

* patients who had primary TKA surgery at six months ago, were diagnosed with preoperative knee OA, and were willing to participate in the research

Exclusion Criteria:

* a previous orthopedic, neurological, or systemic disease that effected walking or standing, body mass index of 40 kg / m2 and over and having any other surgery on the same limb that effected walking.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-01-02 (Actual); Primary Completion 2023-02-12 (Actual); Study Completion 2023-02-12 (Actual)

PRIMARY OUTCOMES:
Short Physical Performance Battery | 1 Hour

SECONDARY OUTCOMES:
TUG | 15 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylul University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ozcan D, Unver B, Karatosun V. Investigation of the validity and reliability of the short physical performance battery in patients undergoing total knee arthroplasty. Physiother Theory Pract. 2025 Feb;41(2):370-376. doi: 10.1080/09593985.2024.2337784. Epub 2024 Apr 1. PMID 38557264